CLINICAL TRIAL: NCT00939510
Title: Phase I/II Study of Lenalidomide (RevlimidTM ) and GM-CSF in Androgen Independent Prostate Cancer
Brief Title: Lenalidomide and GM-CSF in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Robert Dreicer MD (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Robert Dreicer MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3805; P30CA043703 (NIH); IRB# 8121 (Other: Cleveland Clinic IRB); RV-PCA-PI-059
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2012-07-12 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; hormone-resistant prostate cancer; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (RevlimidTM ) and GM-CSF (Experimental)
  Interventions: Biological: sargramostim; Drug: lenalidomide; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: sargramostim — All patients will receive GM-CSF at a dose of 250 mcg subcutaneously on Mondays, Wednesdays and Fridays every week. No dose escalation or de-escalations will be made to GM-CSF.
  Other Names: GM-CSF
Drug: lenalidomide — Lenalidomide will be administered at 25 mg/day orally on days 1-21 of a 28-day cycle. Initially 6 patients will be entered at the 25 mg/day level. If 0 or 1 patients have a dose limiting toxicity, then the 25 mg lenalidomide + GM-CSF 250 mcg subcutaneously on Mondays, Wednesdays and Fridays every week will be accepted as the phase II dose.
Other: laboratory biomarker analysis — Prior to the initiation of each cycle of therapy for the first 3 cycles, and at discontinuation from study blood will be collected for assessments of a prostate cancer specific immune response.

SUMMARY:
RATIONALE: Lenalidomide may stop the growth of prostate cancer by blocking blood flow to the tumor. GM-CSF may stimulate the immune system in different ways and stop tumor cells from growing. Giving lenalidomide together with GM-CSF may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of lenalidomide when given together with GM-CSF and to see how well it works in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Establish the safety of a predetermined target dose or, if the target dose is not tolerable, find the maximum tolerated dose of lenalidomide when administered in combination with sargramostim in patients with androgen-independent prostate cancer.
* Evaluate the preliminary efficacy of this regimen to ascertain whether additional study of lenalidomide is warranted in patients with androgen-independent prostate cancer.
* Evaluate the safety of this regimen in these patients.
* Describe the effects of this regimen on serum cytokines (e.g., TNF-α, bFGF, sIL2R, IL-8, and IL-12) and on serum VEGF levels.
* Assess the co-stimulatory effects of this regimen on CD4+, CD8+, CD83, and CD86 cells.

OUTLINE: This is a phase I, dose-escalation study of lenalidomide followed by a phase II study.

Patients receive oral lenalidomide on days 1-21 and sargramostim subcutaneously on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for correlative biomarker and immunological laboratory studies.

After completion of study therapy, patients are followed up at 30 days and then every 3 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Androgen-independent disease

  * Testosterone ≤ 50 ng/mL

    * Is currently receiving luteinizing hormone-releasing hormone agonists as maintenance or has undergone prior orchiectomy for testosterone suppression
* Progressive disease, as defined by ≥ 1 of the following:

  * Clinical or radiographic evidence of metastases that have progressed irrespective of PSA changes
  * Asymptomatic (non-opioid requiring) bone-only metastatic disease with a rising PSA on separate measurements ≥ 1 week apart

    * No symptomatic bone metastases
  * Biochemical progression (PSA-only disease), defined as having an absolute PSA value of ≥ 2.0 ng/mL on 3 separate measurements ≥ 2 weeks apart with a PSA doubling time of ≤ 10 months
* No evidence of CNS (brain or leptomeningeal) metastases or pleural and/or pericardial effusions

PATIENT CHARACTERISTICS:

* ECOG performance status of 0-1
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Serum creatinine ≤ 2.0 mg/dL
* AST < 3 times normal
* Bilirubin < 1.5 mg/dL
* PT and PTT normal
* Calcium normal
* Fertile patients must use effective contraception during and for ≥ 28 days after completion of study therapy
* Agrees to abstain from donating blood, semen, or sperm during and for ≥ 28 days after completion of study therapy
* No pre-existing peripheral neuropathy > grade 1
* No active unresolved infection
* No known contraindication to lenalidomide or sargramostim
* No other malignancies within the past 5 years, except for curatively treated basal cell or squamous cell carcinoma of the skin or stage Ta transitional cell carcinoma of the bladder

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy for metastatic prostate cancer
* More than 1 year since prior adjuvant and/or neoadjuvant therapy
* More than 4 weeks since prior flutamide (6 weeks for other antiandrogens)
* No prior thalidomide or lenalidomide
* At least 4 weeks since prior surgery or external-beam radiotherapy and recovered
* At least 6 weeks since prior radiopharmaceutical therapy, including samarium-153 or strontium-89, and recovered
* No initiation of bisphosphonate therapy within 1 month before and during study therapy

  * Patients on stable doses of bisphosphonates who show subsequent tumor progression may continue to receive bisphosphonates
* Concurrent daily aspirin for the prevention of thrombotic events required

  * Patients intolerant to aspirin may receive low-dose warfarin as prophylaxis
* No other concurrent investigational agents
* No other concurrent anticancer therapy, including radiotherapy or thalidomide

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-07; Primary Completion 2009-10 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dreicer, MD, FACP, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from November 2005 to April 2009 from medical clinic
Groups:
- Lenalidomide (Revlimid) and Sargramostim (GM-CSF): Sargramostim (GM-CSF) was administered at a dose of 250ug/m2 administered subcutaneously three times weekly every week. No dose escalations or de-escalations of GM-CSF were made. Lenalidomide was administered orally at 25 mg/day on days 1-21 of a 28-day cycle.
Period: Overall Study
Arm/Group | Lenalidomide (Revlimid) and Sargramostim (GM-CSF)
Started | 32
Completed | 31
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide (Revlimid) and Sargramostim (GM-CSF)
Number analyzed (Participants) | 32
Age Continuous [Mean (Standard Deviation); unit: years] | 68.7 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 27
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a PSA Response
Description: Number of patients with a PSA Response defined as a PSA decline greater or equal to 50% compared with baseline value.
Time Frame: reevaluated for response every eight weeks
Population: All patients that received treatment.
Measure: Number; unit: participants
Arm/Group | Lenalidomide (Revlimid) and Sargramostim (GM-CSF)
Number analyzed (Participants) | 31
participants
  PSA response | 4
  PSA no response | 27

2. Secondary Outcome: Number of Patients With Statistically Significant Change in Immune Response From Baseline to End of Study
Description: The change in mean T cell immunohistochemical markers and dendritic cells over time will be evaluated using analysis of variance methods for repeated measures with additional main factors included in the analysis for subset comparisons. The pattern of immune response will be evaluated based upon overall clinical response using these same techniques.
Time Frame: every 28 days for first 3 cycles, end of study
Population: All patients that received treatment
Measure: Number; unit: participants
Arm/Group | Lenalidomide (Revlimid) and Sargramostim (GM-CSF)
Number analyzed (Participants) | 31
participants | 0

3. Primary Outcome: RECIST-defined Measurable Disease
Description: Patients who have a response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) by RECIST criteria. To be assigned a status of PR or CR, changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 4 weeks after the criteria for response are first met. In the case of SD, follow-up measurements must have met the SD criteria at least once after study entry at a minimum interval of 6-8 weeks
Time Frame: every 8 weeks and at end of treatment
Population: 12 patients had RECIST-defined measurable disease. One patient came off study early for toxicity and therefore was not evaluable.
Measure: Number; unit: participants
Arm/Group | Lenalidomide (Revlimid) and Sargramostim (GM-CSF)
Number analyzed (Participants) | 11
participants
  Number of patients with stable disease (SD) | 4
  Number of patients with partial response (PR) | 2
  Number of patients with progressive disease | 5

ADVERSE EVENTS:
Time Frame: Patients followed for adverse events while on study over a three year period.
Arm/Group | Lenalidomide (Revlimid) and Sargramostim (GM-CSF)
Serious Adverse Events (participants affected / at risk) | 5/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (Revlimid) and Sargramostim (GM-CSF) (N=31)
Deep Venous Thrombosis (DVT)/Embolism (Cardiac disorders) | 1
Elevated Lactate dehydrogenase (LDH) (Investigations) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (Revlimid) and Sargramostim (GM-CSF) (N=31)
Anemia (Blood and lymphatic system disorders) | 15
Constipation (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 9
Elevated Lactate dehydrogenase (LDH) (Investigations) | 5
Fatigue (General disorders) | 22
Hypocalcemia (Metabolism and nutrition disorders) | 7
Injection site reactions (General disorders) | 17
Leukopenia (Blood and lymphatic system disorders) | 11
Lymphopenia (Investigations) | 12
Nausea/Vomiting (Gastrointestinal disorders) | 11
Neutropenia (Cardiac disorders) | 12
Skin (dryness, rash, pruritus) (Skin and subcutaneous tissue disorders) | 16
Taste Alterations (Nervous system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes